CLINICAL TRIAL: NCT03430583
Title: Imaging and Biomarker Evaluation of Hepatic Stiffness in Children Enrolled in the Fontan Udenafil Exercise Longitudinal Study
Brief Title: Evaluation of Fontan-associated Hepatic Stiffness and the Efficacy of Udenafil in Reducing Liver Stiffness
Acronym: FALD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mezzion Pharma Co. Ltd (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHN-Udenafil-04; U01HL068270 (NIH)
Record Dates: First submitted 2018-01-22; First posted 2018-02-13 (Actual); Results first posted 2025-09-18 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Single Ventricle Heart Disease
Keywords: Fontan; Ultrasound Shear Wave Elastography; Magnetic Resonance Imaging Elastography
MeSH Terms: interventions — udenafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Udenafil Continuation (U+) (Experimental): Subjects who were receiving Udenafil 87.5 mg BID in FUEL study prior to enrolling to this study (FALD).
  Interventions: Drug: Udenafil
- Udenafil Naive (U-) (Experimental): Subjects who were receiving Placebo BID in FUEL study prior to enrolling to this study (FALD).
  Interventions: Drug: Udenafil

INTERVENTIONS:
Drug: Udenafil — Open-label extension with Udenafil 87.5 mg BID treatment for 52 weeks.

SUMMARY:
A study to evaluate the efficacy of MZ101 therapy in reducing liver stiffness.

DETAILED DESCRIPTION:
This is open-label, long-term prospective study in a cohort of Fontan subjects taking drug daily for one year. The study will determine the scope of hepatic stiffness in the cohort by ultrasound and magnetic resonance imaging elastography and evaluate MZ101 pharmacotherapy as a potentially efficacious treatment to reduce liver stiffness.

ELIGIBILITY:
Inclusion Criteria:

1. Enrollment in on-going Phase 3 Open-Label Safety Study
2. Informed assent from subject, informed consent from parent/legal guardian as appropriate

Exclusion Criteria:

1. Non-enrollment in the on-going Phase 3 Open-Label Study
2. Subjects with contra-indications for MRI (these subjects will be excluded from the MRI component of this study)
3. Other exclusionary criteria will match those used for the Open-Label Safety Study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Goldberg, MD, Principal Investigator — Children's Hospital of Philadelphia; Kurt R Schumacher, MD, Principal Investigator — University of Michigan Congenital Heart Center/C.S. Mott Children's Hospital
Locations (17):
- United States (16):
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Cardiac Center/Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Children's Mercy Hospital, Kansas City, Kansas
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan Congenital Heart Center, Ann Arbor, Michigan
  - Children's Mercy Hospital Kansas City, Kansas City, Missouri
  - University of Nebraska Children's Hospital and Medical Center, Omaha, Nebraska
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Medical Hospital/Dept. of Pediatric Cardiology, Salt Lake City, Utah
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Udenafil Continuation (U+): Treatment subgroup previously exposed to Udenafil
- Udenafil Naive (U-): Treatment subgroup naive to Udenafil
Period: Overall Study
Arm/Group | Udenafil Continuation (U+) | Udenafil Naive (U-)
Started | 36 | 52
Completed | 33 | 45
Not Completed | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Udenafil Continuation (U+): Subset of subjects on Open-label extension study with Udenafil 87.5 mg BID treatment for 52 weeks, who received active Udenafil 87.5 mg BID treatment in FUEL study prior to enrolling to this study (FALD).
- Udenafil Naive (-): Subset of subjects on Open-label extension study with Udenafil 87.5 mg BID treatment for 52 weeks, who received Placebo BID treatment in FUEL study prior to enrolling to this study (FALD).
- Total: Total of all reporting groups
Arm/Group | Udenafil Continuation (U+) | Udenafil Naive (-) | Total
Number analyzed (Participants) | 36 | 52 | 88
Age, Customized [Mean (Standard Deviation); unit: years] | 15.80 (1.992) | 15.16 (1.961) | 15.4 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 19 | 32
  Male | 23 | 33 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 32 | 48 | 80
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 32 | 43 | 75
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter squared] | 21.9 (4.552) | 21.4 (4.174) | 21.6 (4.314)
Height [Mean (Standard Deviation); unit: cm] | 162.08 (10.277) | 164.89 (8.936) | 163.74 (9.552)
Weight [Mean (Standard Deviation); unit: Kg] | 57.48 (13.078) | 58.42 (13.238) | 58.03 (13.105)
Liver Stiffness by Ultrasound Shear Wave Elastography (USWE) [Mean (Standard Deviation); unit: meters/sec] — Baseline liver stiffness was measured in subjects at the start of the study by Ultrasound Shear Wave Elastography (USWE) (meters/second). Population: Baseline results presented for subjects who have data at 52 weeks (i.e., paired-data points).
  meters/sec
    number analyzed (Participants) | 33 | 42 | 75
    (all) | 1.91 (0.380) | 2.02 (0.450) | 1.97 (0.422)
Liver Stiffness by Magnetic Resonance Elastography (MRE) [Mean (Standard Deviation); unit: KiloPascal (kPa)] — Baseline liver stiffness was measured in subjects at the start of the study by Magnetic Resonance Elastography (kilopascal; kPa). Population: Baseline results presented for subjects who have data at 52 weeks (i.e., paired-data points).
  KiloPascal (kPa)
    number analyzed (Participants) | 21 | 17 | 38
    (all) | 5.26 (0.927) | 5.26 (1.453) | 5.26 (1.173)
Enhanced Liver Fibrosis (ELF) [Mean (Standard Deviation); unit: score on a scale] — ELF score is based on the serum levels of hyaluronic acid (HA), amino-terminal propeptide of type III collagen (PIIINP), and tissue inhibitor of metalloproteinase-1 (TIMP-1), and calculated using the following formula: ELF score= 2.494+0.846 In(CHA)+0.391 In(CPIIINP)+0.391 In(CTIMP-1). The normal range in healthy subjects ≤20 years of age is 6.9 - 8.8. Correlations between ELF and the degree of liver fibrosis have not been established in patients with Fontan circulation, however, a decrease in ELF score is associated with improved liver health in other disease states. Population: Baseline results presented for subjects who have data at 52 weeks (i.e., paired-data points).
  score on a scale
    number analyzed (Participants) | 32 | 42 | 74
    (all) | 10.58 (0.915) | 10.45 (0.853) | 10.50 (0.877)
Brain Natriuretic Peptide (BNP) [Mean (Standard Deviation); unit: pg/ml] — Level of Brain Natriuretic Peptide (BNP) was measured in study subjects at baseline. Population: Baseline results presented for subjects who have data at 52 weeks (i.e., paired-data points).
  pg/ml
    number analyzed (Participants) | 32 | 44 | 76
    (all) | 16.89 (13.726) | 17.20 (13.428) | 17.07 (13.464)

OUTCOME MEASURES:

1. Primary Outcome: Effect of Udenafil 87.5 mg BID Treatment on Liver Stiffness in Udenafil Continuation and Naive Groups After 52 Weeks, as Determined by Ultrasound Shear Wave Elastography
Description: Liver stiffness was measured at baseline and 52 weeks using Ultrasound Shear Wave Elastography (USWE) separately in Udenafil Continuation (U+) and Udenafil Naive (U-) groups. A decrease in value indicates a decrease in liver stiffness.
Time Frame: 52 weeks
Population: Only participants with paired data points were included in the analysis population.
Measure: Mean (Standard Deviation); unit: meters per second
Groups:
- Total Udenafil: Total number of subjects exposed to Udenafil treatment during this open-label extension study.
Arm/Group | Udenafil Continuation (U+) | Udenafil Naive (U-) | Total Udenafil
Number analyzed (Participants) | 33 | 42 | 75
meters per second
  Baseline | 1.91 (0.380) | 2.02 (0.450) | 1.97 (0.422)
  Week 52 | 1.86 (0.288) | 1.96 (0.349) | 1.92 (0.325)

2. Primary Outcome: Effect of Udenafil 87.5 mg BID Treatment on Liver Stiffness in Udenafil Continuation and Naive Groups After 52 Weeks, as Determined by Magnetic Resonance Elastography
Description: Liver stiffness was measured at baseline and 52 weeks using Magnetic Resonance Elastography (MRE) separately in Udenafil Continuation (U+) and Udenafil Naive (U-) groups. A decrease in value indicates a decrease in liver stiffness.
Time Frame: 52 weeks
Population: Only participants with paired data points were included in the analysis population.
Measure: Mean (Standard Deviation); unit: kiloPascal (kPa)
Groups:
- Udenafil Continuation (U+): Treatment subgroup exposed to Udenafil
Arm/Group | Udenafil Continuation (U+) | Udenafil Naive (U-) | Total Udenafil
Number analyzed (Participants) | 21 | 17 | 38
kiloPascal (kPa)
  Baseline | 5.26 (0.927) | 5.26 (1.453) | 5.26 (1.173)
  Week 52 | 4.95 (1.080) | 5.50 (1.550) | 5.20 (1.322)

3. Secondary Outcome: Effect of Udenafil 87.5 mg BID on Enhanced Liver Fibrosis (ELF) Score After 52 Weeks of Treatment
Description: Overall ELF score. ELF score is based on the serum levels of hyaluronic acid (HA), amino-terminal propeptide of type III collagen (PIIINP), and tissue inhibitor of metalloproteinase-1 (TIMP-1), and calculated using the following formula: ELF score= 2.494+0.846 In(CHA)+0.391 In(CPIIINP)+0.391 In(CTIMP-1). The levels of each component were as assessed individually and as part of the calculated ELF score as continuous variables. The normal range in healthy subjects ≤20 years of age is 6.9 - 8.8. Correlations between ELF and the degree of liver fibrosis have not been established in patients with Fontan circulation, however, a decrease in ELF score is associated with improved liver health in other disease states.
Time Frame: 52 weeks
Population: Only participants with paired data points were included in the analysis population.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Udenafil Continuation (U+): Patient subgroup previously exposed to Udenafil
- Udenafil Naive (U-): Patient subgroup previously naive to Udenafil
Arm/Group | Udenafil Continuation (U+) | Udenafil Naive (U-) | Total Udenafil
Number analyzed (Participants) | 32 | 42 | 74
score on a scale
  Baseline | 10.58 (0.915) | 10.45 (0.853) | 10.50 (0.877)
  Week 52 | 9.72 (0.818) | 9.79 (0.750) | 9.76 (0.776)

4. Secondary Outcome: Effect of Udenafil 87.5 mg BID on Brain Natriuretic Peptide After 52 Weeks of Treatment
Description: Brain Natriuretic Peptide (BNP) was measured at baseline and 52 weeks of treatment. BNP is a biomarker of overall cardiac function across a variety of disease states. A decrease in value is associated with improved cardiac function.
Time Frame: 52 weeks
Population: Only participants with paired data points were included in the analysis population.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Udenafil Continuation (U+) | Udenafil Naive (U-) | Total Udenafil
Number analyzed (Participants) | 32 | 44 | 76
pg/ml
  Baseline | 16.89 (13.726) | 17.20 (13.428) | 17.07 (13.464)
  Week 52 | 20.31 (18.336) | 20.78 (19.165) | 20.59 (18.698)

ADVERSE EVENTS:
Time Frame: Not applicable, as all safety information was collected in the Study PHN-Udenafil-03 (parent study) and will be reported as part of the results from that study. All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed as part of Study PHN-Udenafil-04.
Groups:
- Udenafil 87.5 mg BID: Open-label extension with Udenafil 87.5 mg BID treatment for 52 weeks.
Arm/Group | Udenafil 87.5 mg BID
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT03430583/Prot_SAP_000.pdf